CLINICAL TRIAL: NCT07159919
Title: The Effect of Insect vs Animal Protein on Post-exercise Skeletal Muscle Anabolic Response and Chronic Adaption to Resistance Training
Brief Title: Insect vs Animal Protein for Building Muscle
Acronym: GAINZ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Collaborators: Aberystwyth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: GAINZ
Record Dates: First submitted 2025-08-26; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Cricket Protein; Whey Protein
Keywords: Insect protein; Sustainable nutrition; Alternative protein; Muscle anabolism; Body composition; Strength; Muscle mass; Resistance training
MeSH Terms: interventions — capsid protein, Cricket paralysis virus; Whey Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cricket protein (Experimental): Group consuming cricket protein
  Interventions: Dietary Supplement: protein supplement
- Whey protein (Active Comparator): Group consuming whey protein
  Interventions: Dietary Supplement: protein supplement

INTERVENTIONS:
Dietary Supplement: protein supplement — Cricket protein incorporated into a whole-food source (dough balls) to be consumed once after an acute bout of resistance exercise and then consumed daily for 12 weeks alongside regular resistance training.
  Other Names: Cricket protein
  Arms: Cricket protein
Dietary Supplement: protein supplement — Whey protein incorporated into a whole-food source (dough balls) to be consumed once after an acute bout of resistance exercise and then consumed daily for 12 weeks alongside regular resistance training.
  Other Names: Whey protein
  Arms: Whey protein

SUMMARY:
This research is being carried out to investigate the potential of insects (crickets) as a sustainable protein source for supporting human muscle tissue by comparing cricket protein to a commonly used animal protein (whey). Insects have been used as protein source for many years in East-Asian and African cultures. More recently the interest in this potential protein source has been growing in Western countries due to the negative environmental impact of producing animal foods and the increased awareness of animal welfare issues in the food chain. Insects are a more sustainable protein source, requiring less land, water and feed, and producing less carbon emissions (greenhouse gases) compared to farming livestock (e.g. cows, pigs, chickens etc.) However, up until now there is no clear evidence that insect-derived protein has the same nutritional properties as animal-derived protein. Recent data from our research group indicates that there appears to be no difference in the digestibility of an insect protein compared to a traditional animal protein amongst younger, middle-aged and older adults. The investigators now want to explore the potential of insect protein to increase muscle mass and strength.

DETAILED DESCRIPTION:
Aims

1. To investigate the impact of insect (cricket) compared to animal (whey) protein on skeletal muscle anabolism (building and repair of muscle tissue) following a bout of resistance exercise.
2. To explore the change in muscle mass and strength following 12 weeks of resistance training whilst consuming cricket or whey protein daily.

Screening

Written informed consent will be taken prior to any procedures being performed. At the screening visit, participants will complete a health questionnaire and basic anthropometric measurements will also be taken (height and weight). The screening session will be conducted by a member of the research team at the University of Surrey physiology lab (Duke of Kent building). If all the inclusion criteria are met, the participant will be invited to join the study. Applicants who don't meet the inclusion criteria will be excluded from the study at this point. Screening data from excluded participants will not be stored, however a summary of how many participants were excluded and for what reasons will be kept for publication purposes. A favourable ethical opinion will be obtained from NHS ethics committee before starting this study. All participants will receive information about the procedures, risks, inconveniences, and benefits of participation from the investigator. Whilst the study does not aim to identify any health irregularities, participants will be informed prior to taking part that if any abnormal health parameter is identified then this will be highlighted to them and they may be advised to follow up with their GP.

Baseline testing

Following the screening visit, participants who have been enrolled onto the study will visit University of Surrey physiology lab to undergo baseline testing. This will begin with a body composition assessment using dual energy x-ray absorptiometry (DEXA), carried out by a trained member of staff who possesses an IR(ME)R certification for body composition scanning. A whole-body DEXA scan will be used to assess lean, fat and bone mass. Participants will then carry out a whole-body dynamic warm up before performing multiple strength tests to assess different indices of muscle strength. This will begin with a countermovement jump to assess explosive strength, followed by an isometric mid-thigh pull to assess maximum force production. This will be followed up by a 1 rep max (1RM) test on the bench press, squat and leg extension to measure upper and lower body maximal strength. The baseline testing will finish with a reps to failure test at 60% of 1RM on the bench press, squat and leg extension. Baseline exercise testing will be carried out by an exercise physiologist.

Phase 1 - Acute anabolic response

Participants will arrive at the lab in the morning after an overnight fast. A baseline venous blood sample (10ml) will be collected via a cannula. A baseline resting muscle biopsy will then be collected from the vastus lateralis of the non-exercise leg using a sterile Bio-Feather™ Semi-Automatic biopsy needle (14 Gauge x 100mm). The biopsy site will be cleaned with a sterile solution and a local anaesthetic (lidocaine) will be injected under the surface of the skin. To avoid any potential confounding effects caused by repeated sampling from the same location, a gap of at least 3cm between sequential biopsies will be maintained. Once the anaesthetic has taken effect, a cannula will be inserted into the muscle. A micro-biopsy needle will then be carefully inserted through the cannula and lowered to the required depth. The needle will be activated, and a small piece of muscle tissue (~20mg) will automatically be collected by the needle, the collection of the sample (from insertion to removal) will take approximately 3 - 5 seconds. Once, complete, the biopsy site will be dressed with a sterile dressing. In total ~60mg muscle tissue will be collected from each biopsy. Muscle tissue will be immediately dissected from any visible adipose or connective tissue and quickly frozen in liquid nitrogen and stored at -80oC until further analysis.

Participants will then perform 5 sets of single-leg resistance exercise using a leg extension machine. They will perform 1 set of 10 reps at 50% of their 1RM determined during the baseline testing visit. Then they will perform 3 sets of 8-10 reps at 80% of 1RM. The final set will also be performed at 80% 1RM but participants will be instructed to keep going until volitional failure if that does not occur after 8-10 reps. A 2-minute rest period will separate each set. This exercise will be overseen by an exercise physiologist.

Immediately following the exercise bout, participants will ingest a baked food product (dough balls) containing 30g of cricket protein (Bugvita, UK) or whey protein (Myprotein, UK). They will be encouraged to consume the food product within a 5-minute period. After ingestion, further blood samples (10ml) will be collected every 20 minutes for the first 60 minutes and then every 30 minutes from 60 - 240 minutes. All participants, regardless of which protein they consume, will also be asked to complete a short taste perception questionnaire to tell us their opinion of how the food product tasted. A further muscle biopsy will be taken from both the resting and exercise leg at 240 minutes after ingestion. In total, 10 blood samples (100ml) and 3 muscle biopsies (~180mg) will be collected during the test visit.

Following the final muscle biopsy, the cannula will be removed, all biopsy dressings will be inspected and then participants will leave the lab. Blood samples will be centrifuged at 1000 x g for 10 minutes at 4oC to separate the plasma, which will then be extracted into aliquots for storage in a -80oC freezer prior to analysis. Muscle tissue samples will be stored in accordance with the Human Tissue Act 2004 in a designated HTA licensed lab at the University of Surrey.

Phase 2 - Chronic training and supplementation

Following phase 1, participants will be randomly assigned to consume 30g of protein from cricket or whey daily for 12 weeks. This will be in the form of the food product used in phase 1. During this time participants will follow a progressive resistance training programme designed to increase muscle mass and strength. Participants will train 3-4 times per week and follow a high protein diet (2g/kg/day) which will be supplemented by the daily intake of cricket or whey protein. The training programme will be designed an exercise physiologist and participants will be instructed not to engage in any other structured exercise during this period.

Participants will be given daily calorie targets based on their estimated total daily energy expenditure to ensure that they are consuming enough energy to grow muscle. A small calorie surplus of 10% will be the daily energy intake target for each participant, given that increasing muscle mass is best achieved in a positive net energy balance. Nutritional targets will be devised by a sports nutritionist.

Participants will be asked to provide a weekly training log via a smartphone app at the beginning, the middle and the end of the 12-week intervention period to ensure that they were performing the required training volume. They will also be asked to provide a 3-day food diary via smartphone app at the beginning, middle and end of the 12-week intervention period to ensure that they were adhering to the nutritional targets set by the research team. The research team will check-in with participants at regular intervals throughout the intervention period either in-person or online to assess progress and tackle any difficulties that participants might be experiencing with the training or dietary targets.

Following the completion of the 12 weeks, participants will return to the University of Surrey physiology lab to repeat the same body composition assessment (DEXA) and strength tests which they performed during the baseline testing visit.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females in general good health (aged 18+)
* BMI between 18.5 and 35 kg/m2
* Weight stable for 3 months (± 2 kg)
* Volunteers must be able and willing to give informed written consent
* Volunteers must be willing to provide blood and muscle tissue samples
* Volunteers must have been resistance training at least 3x per week for a minimum of 2 years
* Volunteers must be willing to follow a resistance training programme and consume a daily protein supplement for 12 weeks
* Not allergic to local anaesthetic

Exclusion Criteria:

* Injury or illness that prevents the adherence to 12 weeks resistance training and protein supplementation
* Those with metabolic conditions such as diabetes
* Those taking nutritional ergogenic aids (e.g. creatine, beta-alanine, sodium bicarbonate, dietary nitrate etc.)
* Those smoking, using nicotine products (e.g., e-cigarettes, patches) or not abstained from these activities for more than 6 months
* Pregnant or lactating (those who become pregnant during this study must notify the researchers immediately and the participant will be removed)
* Volunteers with a habitual caffeine intake >400 mg/day (more than 5 cups standard coffee)
* Drug or alcohol abuse in the last 2 years
* Those who are taking performance enhancing drugs (PEDs) or have previously taken PEDs in the previous 10 years
* Those who do not refrain from alcohol, caffeine containing drinks (e.g., coffee, coca cola, tea, Red Bull) and strenuous exercise 12 hours before the phase 1 visit
* Those with food allergies
* Those following weight loss diets
* Those who are vegan, vegetarian or refrain from dairy/egg consumption

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Anabolic signalling | From baseline measurement to 6 hours later
  Changes in mTORC1 signalling in skeletal muscle from baseline to post-prandial following cricket or whey protein ingestion after exercise
Muscle mass | From baseline measures at enrolment to the end of the training and supplementation period at 12 weeks
  Changes in lean mass following 12 weeks of daily consumption of cricket or whey protein in conjunction with regular resistance training
Muscle strength | From baseline measures at enrolment to the end of the training and supplementation period at 12 weeks
  Changes in muscular strength following 12 weeks of daily consumption of cricket or whey protein in conjunction with regular resistance training

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Manders, PhD, Principal Investigator — University of Surrey
Locations (1):
- University of Surrey, Stag Hill Campus, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD will only be shared amongst the researchers involved in this study.

REFERENCES:
- [Background] Aragon, A., Schoenfeld, B. Magnitude and Composition of the Energy Surplus for Maximizing Muscle Hypertrophy: Implications for Bodybuilding and Physique Athletes. Strength and Conditioning Journal 42(5):p 79-86, October 2020.
- See also: Related Info — https://journals.lww.com/nsca-scj/abstract/2020/10000/magnitude_and_composition_of_the_energy_surplus.9.aspx